CLINICAL TRIAL: NCT05303376
Title: A Randomized, Double-blind, Placebo-Controlled, Escalating Single Dose, Phase 1 & Phase 2 Study to Evaluate the Safety and Efficacy of Inhaled IBIO123 in Participants With Severe COVID-19 Illness
Brief Title: Phase 1&2 Study to Evaluate the Safety & Efficacy of Inhaled IBIO123 in Severe COVID-19 Illness
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Immune Biosolutions Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IBIO-INH-002
Record Dates: First submitted 2022-03-24; First posted 2022-03-31 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Monoclonal antibodies; Inhalation; IBIO; IBIO123; Severe; Hospitalized
MeSH Terms: conditions — COVID-19; Respiratory Aspiration; Lymphoma, Follicular | interventions — IBIO123

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental)
  Interventions: Biological: IBIO123
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: IBIO123 — 5 or 10 mg
  Arms: Active
Other: Placebo — matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 and phase 2, adaptive, placebo-controlled, double-blind, randomized single-dose study in participants with Severe COVID-19 illness.

DETAILED DESCRIPTION:
In Phase 1, in hospital in a continuous observation setting the first cohort will recruit a total of 8 participants who will receive a single inhaled administration of the study treatment. This cohort will consist of 6 participants on active treatment at a dose of 5mg (0.5cc) of IBIO123 and 2 participants on placebo (0.5cc). Participants will be followed for a total duration of 7 days which is greater than 5 expected half-lives of the study drug in lungs. Therefore, after 7 days, negligible amount of the study drug should remain in the lungs of participants. Safety data will be collected and reviewed by a Data Monitoring Committee (DMC). If no stopping rules have been met, the DMC will recommend the dosing of the second cohort at the expected therapeutic dose of 10mg. If stopping rules have been met the DMC will recommend the termination of the study.

The second cohort will be recruited in hospital in continuous observation setting and recruit a total of 8 participants who will receive a single inhaled administration of the study treatment. This cohort will consist of 6 participants on active treatment at a dose of 10mg of IBIO123 (1 cc) and 2 participants on placebo (1 cc).

Participants will be followed for a total duration of 7 days which is greater than 5 expected half-lives of the study drug in lungs. Therefore, after 7 days, negligible amount of the study drug should remain in the lungs of participants. Safety data will be collected and reviewed by a Data Monitoring Committee (DMC). If no stopping rules have been met the DMC will recommend the phase 2 dose of 10mg. If stopping rules have been met the DMC will recommend a phase 2 dose of 5 mg.

In Phase 2, in the lead-in portion of the phase 2, the DMC will meet 7 days after the first 9 subjects (3 Placebo and 6 Active) have completed their day 7 visit to review safety information of these subjects that have been dosed with 10mg of IBIO123 on Days 1 and 3. If this dose regimen is deemed safe by the DMC, the phase 2 study enrolment will pursue and be completed at 10mg on Day 1 and 10 mg on Day 3. If stopping rules were obtained during the Safety review, the study enrolment will be pursued with a single dose of 10mg of IBIO 123 on Day 1.

ELIGIBILITY:
Inclusion Criteria:

Age

1. Are ≥18 years of age at the time of randomization

   Disease Characteristics
2. Are currently hospitalized since less or equal than 3 days for COVID-19 respiratory illness
3. Must have a positive SARS-CoV-2 viral infection determination prior to randomisation. For the phase 2 portion of the study only, the test must be performed within 24 hours before randomisation. Test can be a PCR or an antigen test originated from the institution or any government approved testing site. If the original test result is greater than 24 hours from randomisation, a rapid antigen must be performed at bedside by the study team to determine eligibility

   Sex
4. Are men or non-pregnant women Reproductive and Contraceptive agreements and guidance is provided in Appendix 2. Contraceptive use by men or women should be consistent with local regulations for those participating in clinical studies.

   Study Procedures
5. Understand and agree to comply with planned study procedures
6. Agree to the collection of nasopharyngeal swabs and venous blood

   Informed Consent
7. The participant or legally authorized representative give signed informed consent

   Exclusion Criteria:

   Medical Conditions
8. COVID-19 onset of symptoms began more than 10 days before randomisation
9. Currently intubated or intubation is planned within the next 24 hours
10. Have known allergies to any of the components used in the formulation of the interventions
11. Suspected or proven serious, active bacterial, fungal, viral, or other infection (besides COVID-19) that in the opinion of the investigator could constitute a risk when taking intervention
12. Have any co-morbidity requiring surgery within <7 days, or that is considered life- threatening within 29 days
13. Have any serious concomitant systemic disease, condition, or disorder that, in the opinion of the investigator, should preclude participation in this study.

    Other Exclusions
14. Have received treatment with a SARS-CoV-2 specific monoclonal antibody
15. Have participated, within the last 30 days, in a clinical study involving an investigational intervention. If the previous investigational intervention has a long half-life, 5 half-lives or 30 days, whichever is longer, should have passed.
16. Are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
17. Are pregnant or breast feeding
18. Are investigator site personnel directly affiliated with this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-06-27 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Phase 1: Characterize the effect of IBIO123 compared to placebo on safety and tolerability | Baseline to Day 7
  • Safety assessments such as AEs and SAEs
Phase 2: Characterize the effect of IBIO123 compared to placebo on SARS-CoV-2 viral load and viral clearance | Baseline to Day 5
  • Change from baseline to Day 5 (± 2 days) in SARS-CoV-2 viral load

SECONDARY OUTCOMES:
Phase 1: Characterize the effect of IBIO123 compared to placebo on SARS-CoV-2 viral load and viral clearance | Baseline to Day 7
  • Change from baseline to Day 7 (± 2 days) in SARS-CoV-2 viral load
Phase 2: Characterize the effect of IBIO123 compared to placebo on COVID-19 clinical progression | Baseline to Day 29
  • Change over time from baseline to Day 29 (± 2 days) in COVID-19 WHO Clinical Progression Scale
Phase 2: Characterize the effect of IBIO123 compared to placebo on overall participant clinical status | Baseline to Day 29
  • Proportion (percentage) of participants who experience these events by Day 29
  * ICU admission
  * intubation
  * Mortality
  * Discharge from Hospitalisation
Phase 2: Characterize the effect of IBIO123 compared to placebo on safety and tolerability | Baseline to Day 29
  • Safety assessments such as AEs and SAEs
Phase 2: Characterize the effect of IBIO123 compared to placebo on length of stay in hospital | Baseline to Day 29
  • Mean duration of hospitalisation and ICU care (days)
Phase 2: Characterize the effect of IBIO123 compared to placebo on oxygen supplementation and ventilation needs | Baseline to Day 29
  Mean duration of oxygen treatment (days) and Incidence of Intubation and Mean duration of Intubation (days)
Phase 2: Characterize the pharmacokinetics of IBIO123 | Days 1, 3, 7 and 29
  IBIO123 mean plasma concentration
Phase 2: Characterize the immunogenicity of IBIO123 | Baseline to Day 29
  Assessment of Anti-drug antibodies of IBIO123 at Day 1 and 29

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Labbe, PhD, Study Director — Immune Biosolutions
Locations (5):
- South Africa (2):
  - JOHESE UNITAS Hospital, Lyttelton, Centurion
  - JOHESE ZAH Hospital, Pretoria, Gauteng
- Ukraine (3):
  - Central City Clinical Hospital of Ivano-Frankivsk City Council, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - City Clinical Hospital #1 of Ivano-Frankivsk City Council, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Hospital №1" of the Zhytomyr City Council, Zhytomyr, Zhytomyr Oblast

IPD SHARING:
Plan to Share IPD: No